CLINICAL TRIAL: NCT03735823
Title: The Role of IL-II in the Development of Autoimmune Response in Multiple Sclerosis
Brief Title: IL-11 in the Development of Multiple Sclerosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Other Study IDs: 080-19000-S31301
Record Dates: First submitted 2018-11-07; First posted 2018-11-08 (Actual); Last update posted 2022-06-06 (Actual); Status verified 2022-06

CONDITIONS: Multiple Sclerosis
Keywords: IL-11 T cell migration
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — Blood and CSF samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention, just collect blood samples and CSF samples — No intervention
  Other Names: No intervention

SUMMARY:
Since the last submission, the investigator have further characterized the potential of IL--11 to induce encephalitogenic CD4+IL--17A+, IL--21+ and GM--CSF+ cells, which upon passive transfer induced severe RREAE with IL--17A+CCR6+ CD4+ cell, neutrophil, CD8+ and B--cell accumulation within the CNS (manuscript submitted for publication). These findings confirmed our hypothesis and further characterization of the IL--11--induced encephalitogenic CD4+ cells will be performed as planned in the grant proposal

DETAILED DESCRIPTION:
Immunomodulatory therapies are most effective when administered early in the course of relapsing remitting multiple sclerosis (RRMS). Therefore, investigators are seeking biomarkers of the autoimmune response to accurately identify patients with clinically isolated syndrome (CIS), the earliest phase of the disease. Investigators' preliminary studies have identified IL--11 as the most significantly increased cytokine in the serum and cerebrospinal fluid (CSF) of CIS patients. Serum IL--11 and IL--17A levels correlate with brain MRI T2 and T1 lesion load and were significantly increased during clinical exacerbations in comparison to disease remissions in untreated RRMS patients. Investigators also found that IL--11 induces Th17 cell differentiation and expansion in CIS patients. Investigators' human studies have identified that CD4+ cells represent the predominant source of IL--11 within the peripheral circulation. In comparison to healthy controls (HCs), IL--11+CD4+ cells from CIS patients were significantly increased in the peripheral circulation and exhibited the highest CCR6 expression (86 %) among CD4+ T cell subsets. This implied their potential for early migration to the CNS. Indeed, IL-11+CD4+ cells were significantly enriched in the CSF of RRMS patients in comparison to their matched blood samples (40.9 vs. 2.3%), with the most prominent increase in the number of IL--17A+IL--11+CD4+ cells. Immunohistochemistry studies of active brain MS lesion biopsy samples revealed an enrichment of IL--11+ cells within CD4+ infiltrating cells, suggesting their important role in the development of inflammatory CNS lesions. Animal studies have confirmed the causal role of IL--11 in the exacerbation of RR experimental autoimmune encephalomyelitis (EAE), where IL--11 increased the number of central nervous system (CNS)--infiltrating IL-17A+CD4+ cells in comparison to control mice with EAE, reflecting IL--11 induction of CCR6 expression in CD4+ cells. IL--11Ra KO mice had an attenuated EAE clinical course and lower serum IL--17A levels, as well as lower numbers of Il--17A+CD4+ cells in the brain and spinal cord inflammatory infiltrates, similar to the IL23p19 KO mice. Administration of mouse anti IL--11R mAb in the preclinical phase of EAE induced a delayed onset and decreased disease severity, with decreased IL--17A serum levels. The objectives of this study are to (1) identify the molecular mechanisms involved in the IL--11--induced migration of CD4+ cell subsets to the CNS, (2) Functionally characterize CSF--enriched IL--11+CD4+ cells in CIS patients, (3) examine the potential of IL--11 to induce encephalitogenic CD4+ cells, and determine the therapeutic effect of anti IL--11R mAb in RREAE.

Specific Aims:

Aim 1. Characterize the IL--11--induced migration of CD4+ cell subsets in CIS patients.

1.A. Identify signaling pathways involved in the IL--11--induced migration of CD4+ cell subsets to the CNS. Investigators will identify IL--11--stimulated signaling pathways mediating expression of CCR6 and adhesion molecules on CD45RO+ cells.

1. B. Determine direct chemotactic effect of IL--11 in CD4+ cell subsets. In vitro migration assays will determine a direct chemotactic effect of IL--11 on the migration of CD4+ cell subsets through the endothelial cell (EC) barrier.

   Aim 2. Identify the transcriptional profile and TCRVb repertoire of CSF--enriched IL--11+CD4+ cells from CIS patients.
2. A. Characterize the phenotype and transcriptional profile of CSF--enriched IL--11+CD4+ cells. Flow cytometry phenotyping and RNA sequencing will be performed on IL--11+CD4+ cells from CSF and matched blood samples.

2.B. Determine the TCRVb repertoire of CSF IL--11+CD4+ cells. Identify whether they can be tracked to the peripheral circulation.

Aim 3. Characterize the role of IL--11 in the induction of encephalitogenic CD4+ cells.

3.A. Determine the capacity of IL--11 to induce encephalitogenic CD4+ cells. In vivo experiments will test the effect of IL--11 on the encephalitogenic capacity of CD4+ cells.

3.B. Determine the efficacy of anti IL--11R mAb in preventing and suppressing RREAE. Mice with RREAE will be treated prior to and during the clinical flare--ups and the remission of the disease. The therapeutic effect of anti IL--11R mAb will be characterized via the clinical response, immunohistochemistry, and flow cytometry studies of CNS infiltrating cells.

ELIGIBILITY:
Inclusion Criteria:

First clinical presentation and at least two central nervous system MRI lesions consistent with demyelinating disease;

Age 18-65 inclusive;

Extended disability status score (EDSS) 1.5-5.5;

No immunomodulatory or immunosuppresive therapy prior to the enrollment in the study.

Exclusion Criteria:

Concomitant infection;

Significant medical and psychiatric condition at the disgression of principal investigator;

Pregnant women;

Children and patients participating in research trials will not be enrolled in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 56 untreated patients with CIS according to the Revised McDonald Diagnostic Criteria and 40 control subjects with no evidence of the inflammatory diseases will be enrolled. Female and male subjects will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 96 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2023-05-31 (Estimated); Study Completion 2023-05-31 (Estimated)

PRIMARY OUTCOMES:
Adhesion marker expression of IL-11 producing CD4 T cells in the CNS and peripheral | baseline
  surface adhesion marker Vla-4,Vla-2 and ICAM-1 expression pattern
Cytokine receptor expression of IL-11 producing CD4 T cells in the CNS and peripheral | baseline
  cytokine receptor IL1R,IL6R,IL23R,IL11RA,IL21R and IL17RA expression pattern
Chemokine receptor expression of IL-11 producing CD4 T cells in the CNS and peripheral | baseline
  chemokine receptor CXCR3,CCR7,CCR6,CCR10 and CCR4 expression
transcription factor expression of IL-11 producing CD4 T cells in the CNS and peripheral | baseline
  transcription factor pstat3, Gata3, Tbet,RORrt and Foxp3 expression pattern

CONTACTS AND LOCATIONS:
Overall Officials: Silva Markovic-Plese, MD PhD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided
Investigators probably share data with other potential collaborators for further research